CLINICAL TRIAL: NCT05430490
Title: Cannabis, HIV and Mental Processing Systems
Acronym: CHAMPS
Status: Recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Rutgers University (Other)
Responsible Party: Sponsor
Other Study IDs: 202107149
Record Dates: First submitted 2022-04-25; First posted 2022-06-24 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: HIV Infections; Cannabis
MeSH Terms: conditions — HIV Infections; Marijuana Abuse | interventions — Neuropsychological Tests; Blood Specimen Collection; Surveys and Questionnaires; Spinal Puncture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood and CSF
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- HIV+ Cannabis User: Persons diagnosed with HIV who identify as using medical or recreational marijuana
  Interventions: Procedure: MRI; Other: NeuroPsychological Testing; Procedure: Blood Draw; Other: Questionnaires; Procedure: Lumbar Puncture
- HIV+ Cannabis Non-User: Persons diagnosed with HIV who identify as not using medical or recreational marijuana
  Interventions: Procedure: MRI; Other: NeuroPsychological Testing; Procedure: Blood Draw; Other: Questionnaires; Procedure: Lumbar Puncture
- HIV- Cannabis User: Persons without HIV who identify as using medical or recreational marijuana
  Interventions: Procedure: MRI; Other: NeuroPsychological Testing; Procedure: Blood Draw; Other: Questionnaires; Procedure: Lumbar Puncture
- HIV- Cannabis Non-User: Persons without HIV who identify as not using medical or recreational marijuana
  Interventions: Procedure: MRI; Other: NeuroPsychological Testing; Procedure: Blood Draw; Other: Questionnaires; Procedure: Lumbar Puncture

INTERVENTIONS:
Procedure: MRI — Multimodal neuroimaging on 3T Prisma Fit MRI
Other: NeuroPsychological Testing — A series of written, verbal, and motor tasks requiring the participant to follow instructions, remember words and numbers, draw objects, and complete timed actions.
Procedure: Blood Draw — Laboratory reports (CMP, CBC, Lipids)
Other: Questionnaires — Life history, current behaviors, and substance use surveys
Procedure: Lumbar Puncture — Optional procedure which involves obtaining cerebral spinal fluid through a needle in the lower back

SUMMARY:
This study employs novel methods to identify key determinants and consequences of concurrent HIV infection and regular cannabis use. This study will acquire extensive phenotype data from peripheral and brain markers of immune activation, brain structure, and neuropsychological performance (NP) in persons living with HIV (PLWH) receiving combination anti-retroviral therapy (cART) (80 regular cannabis users and 80 non-users) and HIV uninfected (HIV-) controls (80 regular cannabis users and 80 non-users). This study will provide key insights into the effects of regular cannabis and HIV on peripheral and brain markers of immune function and NP in PLWH and HIV- controls. These insights are critical for cure strategies and ongoing HIV treatment initiatives.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be 18-70 years old.
2. PLWH must have documented HIV infection for approximately 1 year, be on a cART regimen for approximately ≥3 months, and be virally well-controlled (< 200 copies/mL).
3. HIV- controls must have confirmed HIV- serostatus.
4. Participants must complete at least 9 years of education.
5. Participants must be able to provide informed consent.
6. Female participants must have a negative pregnancy test or written documentation of tubal ligation, hysterectomy, post-menopausal status, etc. and cannot be breastfeeding.
7. Participants should have no contraindications to an MRI scan.
8. Participants should be willing to have cannabis use history confirmed via clinical interview and urine analysis .
9. All inclusion criteria at PI discretion.

Exclusion Criteria:

1. History of neurological disorder (e.g., stroke, head injury with loss of consciousness for >5 minutes, developmental learning disability, etc.).
2. Uncontrolled major affective disorder; history of bipolar disorder or schizophrenia. Major depression controlled with no hospitalizations or suicidal ideation in the past year is allowed.
3. Current substance use disorder (SUD) as defined by DSM-5 criteria besides cannabis use disorder (CUD) (though a past SUD > 1 year before the time of study enrolment will be allowed).
4. currently prescribed anti-coagulants (only exclusionary if participant will engage in optional LP).
5. an allergy to lidocaine or similar anesthetic (only exclusionary if participant will engage in optional LP).
6. a history of a bleeding disorder (only exclusionary if participant will engage in optional LP).
7. claustrophobia or a pacemaker that would prevent magnetic resonance imaging (MRI) scanning.
8. all exclusion criteria at PI discretion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 160 PLWH (80 regular cannabis users and 80 non-users) and 160 demographically similar healthy HIV- controls (80 regular cannabis users and 80 non-users) may undergo multimodal neuroimaging, immunophenotyping (including blood and cerebrospinal fluid), and neuropsychological testing to address the specific aims.
Sampling Method: Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2022-03-23 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Effect of cannabis use on peripheral and brain immune activation and inflammation in virally controlled PLWH on cART. | Years 1-5
  Validated plasma and cerebrospinal fluid (CSF) markers of immune health and inflammation (e.g., CD14, CD16, Neopterin, etc.), as well as novel neuroimaging methods of neuro-inflammation (e.g., DTI & DBSI, 3T MRI) will be used to evaluate brain inflammation.

SECONDARY OUTCOMES:
Effect of cannabis use on cognitive performance and brain structure in both PLWH/CB+ and CON/CB+. | Years 1-5
  Neuropsychological assessment results will be normed and converted into Z scores for comparison with brain volumes calculated from the 3T.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Washington University School of Medicine, St Louis, Missouri
  - Rutgers University, Newark, New Jersey

IPD SHARING:
Plan to Share IPD: No